CLINICAL TRIAL: NCT07371598
Title: Impact of Royal Ancient Oats™ on Glycemic Response and Digestive Enzymes
Brief Title: Royal Ancient Oats™ Study
Acronym: RAO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Standard Process Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: SP027
Record Dates: First submitted 2026-01-13; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants; Healthy Glucose
Keywords: healthy glucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Order of receiving muffins differs (Experimental): A: Order of receiving muffins differs
  Interventions: Dietary Supplement: Royal Ancient Oat Flour™
- B: Order of receiving muffins differs (Experimental): B: Order of receiving muffins differs
  Interventions: Dietary Supplement: Royal Ancient Oat Flour™

INTERVENTIONS:
Dietary Supplement: Royal Ancient Oat Flour™ — muffins made with Royal Ancient Oat Flour™

SUMMARY:
Evaluating the effects of high avenanthramide ancient oat (Royal Ancient Oats™) muffins versus conventional oat muffins in regard to glycemic control.

DETAILED DESCRIPTION:
This study is a randomized, two-period crossover trial with a run-in control baseline and repeated measures, designed to evaluate the effects of high avenanthramide ancient oat (Royal Ancient Oats™) muffins versus conventional oat muffins on glycemic control and related metabolic parameters. A total of 38 non-diabetic adults (HbA1c < 5.7%), who are either overweight (BMI 25-29.9) or obese (BMI ≥ 30) will start with a repeated measures baseline using regular flour (white wheat) muffins for three consecutive days. Following this, participants will be divided into two groups: 19 in the conventional oat muffin group and 19 in the Royal Ancient Oats™ muffin group. This sample size provides 90% power to detect a difference in AUC of at least 20% between treatments, with a two-sided alpha of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Non-diabetic (HbA1c<5.7%) adults both men and women between the ages of 35-65 years with body mass index (BMI) ranging from 25 to 30 kg/m2
* Participants who meet the inclusion criteria will be screened prior to starting the study and must be able to adhere to the requirements of the study.
* Willing to comply with study procedures and supplement regimens.
* Providing consent to participate in the study.
* Willing to limit/minimize foods that are rich sources of fiber and high carb content.
* Participants should avoid taking any non-prescription/over-the-counter medications or nutritional supplements that could influence glycemic response. This includes vitamins, herbal supplements, and any medications affecting metabolism. Examples include probiotics and prebiotics, vit D, vit B12, Ginseng, fenugreek, weight loss supplements like green tea extract and Garcinia cambogia, fiber supplements like inulin and Psyllium husk. If participants need to make any changes due to health reasons, they should consult with the study coordinator before doing so.

Exclusion Criteria:

* Participants who have experienced weight loss or gain exceeding 5% of their body weight in the past 3 months, including those involved in any weight loss or weight gain programs through diet and/or lifestyle changes.
* Participants currently taking medications that could alter metabolism, such as weight loss medications, anti-hypertensive drugs, or lipid-lowering medications.
* Participants with any chronic metabolic diseases, including diabetes, or those using supplements other than a daily multivitamin.
* Pregnant or lactating women will be excluded from the study.
* Participants who use tobacco products.
* Participants who are unwilling to limit or minimize foods that are rich sources of fiber and high carbohydrate content.
* Excessive alcohol consumption (e.g., more than two drinks per day for men and more than one drink per day for women)
* Inconsistency in recent or planned changes in non-prescription/over-the-counter medications or nutritional supplements affecting glycemic response, including vitamins (e.g., Vitamin D, Vitamin B12), herbal supplements (e.g., Ginseng, Fenugreek), weight loss supplements (e.g., green tea extract, Garcinia cambogia), fiber supplements (e.g., inulin, psyllium husk), and probiotics/prebiotics.
* Inability or unwillingness to maintain the current regimen of these medications and supplements throughout the study period without consulting the study coordinator.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
To compare the effect of consuming high avenanthramide Royal Ancient Oats™ muffins or conventional oat muffins versus white wheat flour muffins on postprandial glycemic response. | 2 weeks
  Area Under the Curve (AUC) for glucose levels over 24 hours, as measured by Continuous Glucose Monitoring (CGM).

SECONDARY OUTCOMES:
To evaluate the effect of Royal Ancient Oats™ on incretin hormone secretion and satiety hormones. | 2 weeks
  Subjective measures of hunger and satiety using Visual Analog Scales (VAS).
To evaluate the effect of Royal Ancient Oats™ on incretin hormone secretion and satiety hormones. | 2 weeks
  Changes in GLP-1 levels (pg/mL)
To evaluate the effect of Royal Ancient Oats™ on incretin hormone secretion and satiety hormones. | 2 weeks
  Changes in leptin (pg/mL)
To evaluate the effect of Royal Ancient Oats™ on incretin hormone secretion and satiety hormones. | 2 weeks
  Changes in adiponectin (ng/mL)
To evaluate the effect of Royal Ancient Oats™ on incretin hormone secretion and satiety hormones. | 2 weeks
  Changes in peptide YY (pg/mL)

OTHER OUTCOMES:
To evaluate changes in weight, waist circumference, and body composition before and after dietary intervention. | 2 weeks
  Changes in body weight (kilograms, kg) measured using a calibrated digital scale (InBody)
To evaluate changes in weight, waist circumference, and body composition before and after dietary intervention. | 2 weeks
  Changes in waist circumference (centimeters, cm) measured using a flexible, non-stretchable measuring tape at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest.
To evaluate changes in weight, waist circumference, and body composition before and after dietary intervention. | 2 weeks
  Changes in body fat percentage (%) as measured by bioelectrical impedance analysis (e.g., InBody).
To evaluate changes in weight, waist circumference, and body composition before and after dietary intervention. | 2 weeks
  Changes in skeletal muscle mass (kg) as measured by bioelectrical impedance analysis (e.g., InBody).
To evaluate changes in weight, waist circumference, and body composition before and after dietary intervention. | 2 weeks
  Changes in visceral fat level (arbitrary units) as measured by bioelectrical impedance analysis (e.g., InBody).

CONTACTS AND LOCATIONS:
Locations (1):
- Standard Process Nutrition Innovation Center, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shehzad A, Rabail R, Munir S, Jan H, Fernández-Lázaro D, Aadil RM. Impact of Oats on Appetite Hormones and Body Weight Management: A Review. Curr Nutr Rep. 2023 Mar;12(1):66-82. doi: 10.1007/s13668-023-00454-3. Epub 2023 Feb 15. PMID: 36790719; PMCID: PMC9930024.
- [Background] Zhouyao H, Malunga LN, Chu YF, Eck P, Ames N, Thandapilly SJ. The inhibition of intestinal glucose absorption by oat-derived avenanthramides. J Food Biochem. 2022 Oct;46(10):e14324. doi: 10.1111/jfbc.14324. Epub 2022 Jul 27. PMID 35892210
- [Background] Chen CY, Milbury PE, Collins FW, Blumberg JB. Avenanthramides are bioavailable and have antioxidant activity in humans after acute consumption of an enriched mixture from oats. J Nutr. 2007 Jun;137(6):1375-82. doi: 10.1093/jn/137.6.1375. PMID 17513394
- [Background] Chen V, Zurbau A, Ahmed A, Khan TA, Au-Yeung F, Chiavaroli L, Blanco Mejia S, Leiter LA, Jenkins DJA, Kendall CWC, Sievenpiper JL. Effect of oats and oat ß-glucan on glycemic control in diabetes: a systematic review and meta-analysis of randomized controlled trials. BMJ Open Diabetes Res Care. 2022 Sep 1;10(5):e002784. doi: 10.1136/bmjdrc-2022-002784. PMCID: PMC9438016.
- [Background] Trainer VL, McPhee JC, Boutelet-Bochan H, Baker C, Scheuer T, Babin D, Demoute JP, Guedin D, Catterall WA. High affinity binding of pyrethroids to the alpha subunit of brain sodium channels. Mol Pharmacol. 1997 Apr;51(4):651-7. doi: 10.1124/mol.51.4.651. PMID 9106631
- [Background] Raguindin PF, Adam Itodo O, Stoyanov J, Dejanovic GM, Gamba M, Asllanaj E, Minder B, Bussler W, Metzger B, Muka T, Glisic M, Kern H. A systematic review of phytochemicals in oat and buckwheat. Food Chem. 2021 Feb 15;338:127982. doi: 10.1016/j.foodchem.2020.127982. Epub 2020 Sep 5. PMID 32950005
- [Background] Williamson V. Patients' liaison group. Br J Gen Pract. 1993 Jul;43(372):308. No abstract available. PMID 8398256
- [Background] Loskutov, I. G., Gnutikov, A. A., Blinova, E. V. & Rodionov, A. V. The Origin and Resource Potential of Wild and Cultivated Species of the Genus of Oats (Avena L.). Russ J Genet 57, 642-661 (2021)
- [Background] Sood, V. K., Sanadya, S. K., Kumar, S., Chand, S. & Kapoor, R. Health benefits of oat (Avena sativa) and nutritional improvement through plant breeding interventions. Crop Pasture Sci 74, 993-1013 (2022).
- [Background] Stewart, D. & McDougall, G. Oat agriculture, cultivation and breeding targets: Implications for human nutrition and health. in British Journal of Nutrition vol. 112 S50-S57 (Cambridge University Press, 2014).
- [Background] Ociepa, T. The oat gene pools - Review about the use of wild species in improving cultivated oat. Journal of Central European Agriculture 20, 251-261 (2019).
- [Background] Sang, S., & Chu, Y. (2017). Whole grain oats, more than just a fiber: Role of unique phytochemicals. Molecular Nutrition & Food Research, 61(7), 1600715.
- [Background] Pearson, R. W., Aldrich, D. G., H Allaway J E Dawson, J. W. & Gardner E G Heyne F L Patterson, C. O. Oats and Oat Improvement. vol. 4 https://acsess.onlinelibrary.wiley.com/doi/ (1952).
- [Background] Coffman, F. A. Oat History, Identification and Classification. (1977).